CLINICAL TRIAL: NCT07087366
Title: Enhanced Recovery After Surgery(ERAS) Pathway Following Gynecological Oncology Surgery in a Tertiary Level Hospital:A Prospective Randomized Controlled Trial
Brief Title: Enhanced Recovery After Surgery(ERAS) Following Gynaecological Oncology Surgery in a Tertiary Level Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, JANNAT FERDOUS, Professor of Department of gynaecological-oncology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1139
Record Dates: First submitted 2025-06-17; First posted 2025-07-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: ERAS; Cancer
Keywords: RCT
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients between the age of 18-70 years, who will diagnosed with cervical tumors, uterine tumors or ovarian tumors, and admitted for surgical management will be eligible for enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERAS group (Experimental): Preoperative:
  * Education
  * No bowel preparation
  * Fasting up to 6 h before surgery
  * Oral carbohydrate solution (50 G in 200 mL water, 2 hours before surgery
  Day of surgery:
  * Insertion of Foley catheter
  * Antiembolic stockings
  * Fluid restriction (4-5 L)
  * 0.2% Bupivacaine during incision closure
  * Sip of water 2 hours later after surgery
  * Postoperative LMWH injection
  * Antiembolic stockings
  * Foley removal as early as possible
  * Drain removal as early as possible
  * Ambulation at morning & continue and encourage ambulation
  * Fluid restriction (1-2 L
  * NSAIDs/ Paracetamol bid for 3 days for analgesia IV PCA (Epidural)
  * Semifluid diet in POD1
  * Soft blended diet in POD2
  Interventions: Procedure: ERAS protocol
- Conventional Group (No Intervention): Before and after Surgery:
  * Bowel preparation
  * Midnight fasting
  * Insertion of Foley catheter
  * Antiembolic stockings
  * Fluid (5-6L)
  * Fluid (2L-3L)
  * Semifluid diet after first flatus
  Post-operative:
  * Use of Narcotic analgesia
  * Prolonged immobilization
  * NPO till bowel sound
  * Prolonged catheterization

INTERVENTIONS:
Procedure: ERAS protocol — Procedure: ERAS protocol
  Arms: ERAS group

SUMMARY:
Enhanced recovery after surgery (ERAS) protocols are multimodal perioperative care pathways designed to achieve early recovery after surgical procedures by maintaining preoperative organ function and reducing the profound stress response following surgery.

The principle of ERAS is to optimize the patient's health before surgery, minimize stress to the body, and restore function to normal rapidly by taking steps before, during, and after surgery, to decrease the length of stay in the hospital, reduce recovery time, prevent complications, readmissions, same day discharge (SDD) and patient's satisfaction.

The aim of this study is to introduce the ERAS recommendations into the management of gynaecological surgical procedures in compared to conventional procedures.

After taking permission from Institutional Review Board (IRB) of BSMMU, the proposed study will be started. After taking informed written consent and matching eligibility criteria, a total 160 patients will be selected in this prospective randomized control study. This study will be conducted in the Department of gynecological oncology, BSMMU for two years from April 2024 to March 2026. There will be two group in this study, patients of Group A will be selected for ERAS protocol from preoperative to postoperative event up to follow up. Patients of Group B will be selected for conventional method. Outcome of both procedure in terms of hospital stay, costs, requirement of analgesia and complications will be compared. Statistical analyses of the results will be obtained by using window-based computer software devised with Statistical Packages for Social Sciences (SPSS-25).

DETAILED DESCRIPTION:
Over 234 million major surgical procedures are performed globally each year and despite advances in surgical and anaesthetic care, morbidity after abdominal surgery is still high. Fasttrack or enhanced recovery after surgery (ERAS) clinical pathways have been proposed to improve the quality of perioperative care with the aim of attenuating the loss of functional capacity and accelerating the recovery process.

The ERAS pathways reduce the delay until full recovery after major abdominal surgery by attenuating surgical stress and maintaining postoperative physiological functions. The implementation of the ERAS pathways has been shown to impact positively in reducing postoperative morbidity, and as a consequence, length of stay in hospital.

The concept of ERAS was first published by Engelman and colleagues in cardiac surgery in 1994. Subsequently, ERAS Society was formed in the early 2000s by a group of European surgeons (ERAS Society guidelines was formed). Early studies were primarily focused on colorectal surgery, and in 2003 (Marx and colleagues) this concept was demonstrated in gynecologic oncology. The first ERAS guidelines in gynecologic oncology were published in 2016. Updated guidelines for ERAS in gynecologic oncology were published in 2019.

Components of ERAS are preoperative, intraoperative and post operative. Pre-operative component includes: Patient education regarding the surgery and the expected post-operative course, ensuring the patient is as healthy as possible prior to surgery through exercise & weight loss, optimal pre-operative fasting guidelines that will allow solid food until 6 hours pre-operatively and intake of clear fluids until 2 hours prior to surgery. A Cochrane review reported that preoperative carbohydrate treatment was associated with reduced post-operative insulin resistance, enhanced return of bowel function, and shorter hospital stay with no effect on post-operative complication rates, length of hospital stay (LOSH) and its related costs. In recent years, several studies have highlighted the impact of the anaesthetic management on postoperative morbidity and mortality.

In view of the evidence that many elements of the ERAS programme published by the ERAS Society in 2009 are of related to anaesthetic care, it is imperative that guidelines on perioperative care include recommendations approved by an interdisciplinary team comprising anaesthesiologists and surgeons.

Most of the ERAS elements have been already discussed extensively, specifically for different types of surgical procedures, as well the quality of evidence supporting each ERAS element. It must be acknowledged that evidence supporting some of the ERAS elements still remains controversial. The historical significance of ERAS has been established since 1990 (REF) in general surgery, orthopaedics and urology. ERAS resulted in increased patient satisfaction, shorter hospital stays, reduced postoperative complications and reduced treatment costs, which contribute to increased hospital productivity.

There are a number of reports in the literature on the implementation of the ERAS programme into the care of gynaecological patients . Minimally invasive surgery is advisable in ERAS protocol in order to reduce surgical complications, wound infections, incidence of deep vein thrombosis and hospital stay.

There is a strong opinion that the majority of gynaecological procedures can be done without mechanical bowel preparation (enema) .

One of the demonstrated advantages of restricting the administration of intravenous fluids to surgical patients is the reduction of pulmonary complications . Another recommendation is the avoidance of opioids, which can cause nausea, vomiting and ileus .

Regarding Health Economics Benefits; Direct medical and indirect non-medical costs were significantly lower in the ERAS group, there was a significant reduction in total hospital stay, intravenous fluid use, complications and duration of epidural use in the ERAS group, The implementation of an ERAS program causes overall cost-saving of roughly $6900 per patient.

The aim of this study is to introduce the ERAS recommendations into the management of gynaecological procedures in our institution.

Rationale of the research:

Optimization of care in the perioperative period is increasingly being recognized as a means of improving outcomes after surgery. This began with the concept of enhanced recovery after surgery (ERAS) which described pre, intra, and post-operative factors to improve patient outcomes after surgery.

Following recommendations are advocated for preoperative preparation while doing major gynaecological oncological surgery: No preoperative mechanical bowel preparation as several studies have shown that oral antibiotics alone compared with no bowel preparation significantly reduced post-operative infectious morbidity including anastomotic leaks. ERAS protocol also recommend that all gynecologic oncology patients who undergo major surgery > 30 min should receive dual VTE mechanical prophylaxis and chemoprophylaxis. Perioperative prophylaxis should begin before the induction of anesthesia Intra-operative component includes use of multimodal and opioid-sparing analgesia, targeting perioperative goal-directed fluid therapy that reduces length of stay & complications in high-risk patients undergoing abdominal surgery . Minimally invasive surgery remains an important tenet of ERAS and is recommended for appropriate patients when long-term oncologic outcomes are similar, where expertise and resources are available .

Post-operative component includes adequate pain control, early mobilization, early oral intake. A regular diet within the first 24 hours after gynecologic/oncology surgery is recommended, High protein diets may be considered, multi-disciplinary post-operative patient follow-up is required. Patient Reported Outcomes, including functional recovery and audit also one of the most important component of ERAS protocol that allow institutions to monitor, understand, and compare functional recovery in a patient-centered fashion.

But the conventional protocol that has been practicing for our patients so far is complicated as it involves preoperative mechanical bowl preparation that stats 3 days prior to surgery, preoperative and post operative use of opioids and more analgesics.

So, the conventional protocol causes more length of hospital stay, patients discomfort and less turn over that ultimately increase hospital cost for the patients.

There are limited study done to evaluate the optimization of ERAS protocol in Bangladesh and no study was performed so far in gynaecological cancer surgery. This study is done to determine the ultimate outcome of gynaecological oncology surgery following ERAS protocol and compare it with the conventional method in BSMMU .

Hypothesis:

The perioperative and post operative in patients undergoing gynaecological cancer surgeries following ERAS protocol is better than that of the conventional method.

Objective:

General objective:

To find out the perioperative and postoperative outcome in patients undergoing gynaecological cancer surgeries following ERAS protocol (Group A) compared with conventional method(Group B).

Specific objectives:

1. To compare the perioperative pain score, day of first flatus, any complications in patients undergoing gynaecological cancer surgeries following ERAS protocol and in patients following conventional protocol.
2. To compare the costs , hospital stay, complications, readmission rate, reoperation rate, postoperative mortality in both the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18-70 years,
* diagnosed case with cervical, uterine or ovarian cancer,
* Admitted for surgical management .

Exclusion Criteria:

* Patients with severe comorbidity, including DM,CRD,CLD
* patients with American Society of Anesthesiologists risk ≥ 4,
* severe organ dysfunction or failure.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
hospital stay | 3 to 4 days
  duration of hospital stay in ERAS group

SECONDARY OUTCOMES:
Day of first flatus | upto 24 hours
  day of first flatus
postoperative nausea and vomiting | upto 24 hours
  frequency of postoperative nausea and vomiting
pain score by the visual analogue scale with score minimum 0 and maximum 10 | upto 48 hours
  pain score from the scale that is higher score indicate worse and lower score indicate good
complications related to the intervention | upto 2 weeks
  yes or no
readmission rate | upto 21days
  readmission rate
mortality rate after the procedure | 5 to 7 days
  postoperative mortality rate and number
Total hospital cost | 3to 4 days
  total hospital cost

CONTACTS AND LOCATIONS:
Overall Officials: JANNAT FERDOUS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Jannat Ferdous, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No